CLINICAL TRIAL: NCT02897518
Title: Comparison Between Imago V-Blade and Glidescope During Endotracheal Intubation: a Feasibility Study
Brief Title: Videolaryngoscopes for Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Maria Vargas, MD, Federico II University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Airway1
Record Dates: First submitted 2016-08-25; First posted 2016-09-13 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Airway Management
Keywords: Videolaryngoscopes; Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endotracheal intubation with Imago V-blade (Experimental): Patients in this arm will receive endotracheal intubation with the Imago V-Blade videolaryngoscopes.
  Interventions: Device: Imago V-Balde
- endotracheal intubation with Glidescope (Active Comparator): Patients in this arm will receive endotracheal intubation with the glidescope videolaryngoscopes.
  Interventions: Device: Glidescope

INTERVENTIONS:
Device: Imago V-Balde — the endotracheal intubation will be performed with videolaryngoscopes (imago V-Blade) according to the user manual
  Arms: endotracheal intubation with Imago V-blade
Device: Glidescope — the endotracheal intubation will be performed with videolaryngoscopes (Glidescope) according to the user manual
  Arms: endotracheal intubation with Glidescope

SUMMARY:
The primary end point of this study is the feasibility of intubation. The secondary end-points are the success to intubate in the first attempt, the intubation time, the Cormack and Lehane score view, the comparison of the intubation difficulty scale (IDS) score and the need for maneuvers to aid the endotracheal intubation comparing Imago V-Blade ® and Glidescope®.

Patients admit to the operation rooms of University of Naples "Federico II" and requiring endotracheal intubation for general anesthesia will be consecutively screened for the presence of predicted difficult airway according Italian guideline. According to this guideline, the presence of one or more of the following parameters may be considered highly predictive of difficult intubation: Mallampati class 3-4, inter-incisor distance < 30 mm, mental-thyroidal distance < 60 mm, large prominence of superior incisors above inferior incisors uncorrectable with jaw-thrust, reduced head and neck motility, and reduced mental-jugular distance. Patients matching more then 1 of the previous criteria stated by Italian guideline will be included in this case controlled study. Patients 1) without criteria for predicted difficult airway; 2) those requiring emergency surgery; 3) aged < 18 years; or 4) declined consent to participate, will be excluded from this study.The primary end-point was the comparison of the intubation difficulty scale (IDS) score. The secondary end-points were the learning curve, the intubation time, the Cormack and Lehane score view, and the need for maneuvers to aid the endotracheal intubation comparing different videolaryngoscopes available in our department. Two anesthesiologists with 10 years of experience in conventional endotracheal intubation and trained for video assisted intubation will perform the maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Mallampati class 3-4
* inter-incisor distance < 30 mm
* mental-thyroidal distance < 60 mm
* large prominence of superior incisors above inferior incisors uncorrectable with jaw-thrust -reduced head and neck motility
* reduced mental-jugular distance.

Exclusion Criteria:

* < 1 criteria for predicted difficult airway
* emergency surgery
* age < 18 years
* declined consent to participate

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
feasibility of endotracheal intubation | within 60 seconds

SECONDARY OUTCOMES:
Success rate of endotracheal intubation using Imago V-Blade compared with Glidescope | wthin 120 seconds
  Time to reach a successful endotracheal intubation from the beginning of indirect laryngoscopy to the confirmation of the intubation with the evaluation of the end-tidal carbon dioxide
Intubation time | wthin 120 seconds
  time to reach endotracheal intubation from the beginning of indirect laryngoscopy to the confirmation of the intubation with the evaluation of the end-tidal carbon dioxide
Cormack and Lehane score view | During endotracheal intubation
use of adjunctive maneuvers to aid the endotracheal intubation | During endotracheal intubation
  the investigators evaluated the necessary maneuvers to aid a successful endotracheal intubation as number of Readjusting patient's head, number of external laryngeal pressure, number of advancement or withdrawal the blade and number of increased lifting force
Intubation difficulty scale score | within 60 seconds
  Time to pass the vocal cord during the successful endotracheal intubation measured from the beginning of indirect laryngoscopy to the confirmation of the intubation with the evaluation of the end-tidal carbon dioxide

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II department of Anesthesia and Critical Care, Naples, Italy, Italy

REFERENCES:
- [Derived] Vargas M, Pastore A, Aloj F, Laffey JG, Servillo G. A comparison of videolaryngoscopes for tracheal intubation in predicted difficult airway: a feasibility study. BMC Anesthesiol. 2017 Feb 20;17(1):25. doi: 10.1186/s12871-017-0318-2. PMID 28219331